CLINICAL TRIAL: NCT00774917
Title: Numen Stent Assessment Using OCT Technique in a Single Center Study
Acronym: NAUTIC
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Biomedical Systems S.p.A. (Industry)
Collaborators: CSC Pharmaceuticals (Industry)
Responsible Party: Univ. Prof. Dr. Helmut-Dietmar Glogar, Universitary Hospital of Wien (Vienna - Austria)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSC-IBS/05-2007
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2009-06-23 (Estimated); Status verified 2009-06

CONDITIONS: Hyperplasia; Restenosis
Keywords: numen; hyperplasia
MeSH Terms: conditions — Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Numen (Experimental)
  Interventions: Device: Numen

INTERVENTIONS:
Device: Numen — Numen Co-Cr coronary stent implant

SUMMARY:
This is a prospective single centre Study designed to assess by OCT the effect of NUMEN cobalt-chromium balloon-expandable stent in inducing neointimal hyperplasia in de novo native coronary lesions of patients with Stable Angina Pectoris or ACS (except STEMI).

A total of 60 consecutive patients will be enrolled in the study. Patients with de novo native coronary artery lesions >10mm and <24mm in length and >2.50mm to <3.50mm in diameter by QCA estimate who meet all eligibility criteria will be enrolled and undergone stent implantation. After stent deployment an OCT imaging will be performed within the treated segment. Patients will be followed at 30 days, 6 months and 12 months post-procedure, with all patients having repeat angiography and OCT at 6 months.

It is anticipated that the total length of the study will be 18 months: 6 months to complete patient enrolment and 12 months for follow-up.

DETAILED DESCRIPTION:
OBJECTIVES

The main objective of this study is to assess the long term influence of NUMEN cobalt-chromium balloon-expandable coronary stent on neointimal hyperplasia in de novo native coronary lesions of patients with Stable Angina Pectoris or Acute Coronary Syndrom (ACS) - except STEMI.

ENDPOINTS

The primary endpoint is the assessment of the development of neointimal hyperplasia by OCT in the stented segment at 6-month follow-up.

Breakdown of secondary endpoints:

Degree of endothelialization of the stent internal wall by OCT at 6 months after stent implantation; Composite of Major Adverse Cardiac Events (MACE) defined as cardiac death, non-fatal myocardial infarction (MI) (Q wave and non-Q wave), emergent bypass surgery, stent thrombosis, or repeat target lesion revascularization at 30 days, 6 months and 12 months post-procedure.

Angiographic binary restenosis (>50% diameter stenosis) 6 months post-procedure.

Target vessel failure at 6 months post-procedure. Device success defined as achievement of a final residual diameter stenosis of <30% (by Quantitative Coronary Angiography (QCA)), using the assigned device only. If QCA is not available, the visual estimate of diameter stenosis is used.

Lesion success defined as the attainment of <30% residual stenosis (by QCA) using any percutaneous method.

Procedure success defined as achievement of a final diameter stenosis of <30% (by QCA) using any percutaneous method, without the occurrence of death, MI, or repeat revascularization of the target lesion during the hospital stay.

Acute (24 hrs post procedure), subacute (up to 30days post procedure) and late (>30days post procedure) thrombosis.

OVERVIEW OF THE STUDY

This is a prospective single centre Study designed to assess by OCT the effect of NUMEN cobalt-chromium balloon-expandable stent in inducing neointimal hyperplasia in de novo native coronary lesions of patients with Stable Angina Pectoris or ACS (except STEMI).

A total of 60 consecutive patients will be enrolled in the study. Patients with de novo native coronary artery lesions >10mm and < 24mm in length and >2.50mm to <3.50mm in diameter by QCA estimate who meet all eligibility criteria will be enrolled and undergone stent implantation. After stent deployment an OCT imaging will be performed within the treated segment. Patients will be followed at 30 days, 6 months and 12 months post-procedure, with all patients having repeat angiography and OCT at 6 months.

It is anticipated that the total length of the study will be 18 months: 6 months to complete patient enrolment and 12 months for follow-up.

ELIGIBILITY:
INCLUSION CRITERIA

Patients must meet all of the following criteria:

1. The patient must be > 18 years of age;
2. Diagnosis of stable angina pectoris as defined by Canadian Cardiovascular Society Classification (CCS I, II, III, IV) or ACS (except STEMI).
3. Treatment of de novo lesion in a major coronary artery in patients with single or two-vessel disease.
4. Target vessel diameter at the lesion site is >2.50mm and <3.50mm in diameter (QCA);
5. Target lesion is >10mm and <24mm in length (visual estimate);
6. Target lesion stenosis is >50% and <100% (visual estimate);
7. Acceptable candidate for coronary artery bypass surgery (CABG);
8. Patient is willing to comply with the specified follow-up evaluation;
9. Patient must provide written informed consent prior to the procedure using a form that is approved by the local Ethics Committee.

EXCLUSION CRITERIA

Patients will be excluded if any of the following conditions apply:

1. multiple lesions in the same vessel;
2. ACS with STEMI (within 48 hours)
3. vessel size < 2.50mm and >3.50mm reference diameter;
4. length of the lesion > 24 mm;
5. unprotected left main coronary disease with >50% stenosis;
6. have an ostial target lesion;
7. have a target lesion in a venous graft;
8. angiographic evidence of thrombus within target lesion;
9. calcified lesion which cannot be successfully predilated;
10. Documented left ventricular ejection fraction >25%;
11. Impaired renal function (creatinine > 3.0 mg/dl) at the time of treatment;
12. Pretreatment with devices other than balloon angioplasty;
13. Prior stent within 5mm of target lesion;
14. Recipient of heart transplant;
15. Known allergies to the following: aspirin, clopidogrel bisulfate (Plavix) and ticlopidine (Ticlid), heparin, cobalt, chromium, or contrast agent (that cannot be managed medically)
16. Recent (6 months) cerebrovascular accidents or intracranial hemorrage
17. Any significant medical condition which in the investigator's opinion may interfere with the patient's optimal participation in the study;
18. Currently participating in an investigational drug or another medical device study;
19. In the investigator's opinion, the lesion is not suitable for stenting.
20. Life expectancy ≤ 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-09 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is the assessment of the development of neointimal hyperplasia by OCT in the stented segment at 6-month follow-up. | 6 months

SECONDARY OUTCOMES:
Endothelialization of the stent internal wall by OCT at 6 months ; (MACE) at 30 days, 6 and 12 months Angiographic binary restenosis at 6m Target vessel failure at 6m. Device, lesion, procedure success. Thrombosis | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Dietmar Glogar, Prof., Principal Investigator — University Hospital of Vienna
Locations (2):
- Austria (2):
  - University Hospital of Vienna, Vienna (Austria), Vienna
  - SMZ-Ost Donauspital, Vienna